CLINICAL TRIAL: NCT06157983
Title: Evaluation of Cascade Screening for Elevated Lipoprotein(a) in Relatives to Patients With Atherosclerotic Coronary Artery Disease
Brief Title: Evaluation of Cascade Screening for Elevated Lipoprotein(a)
Acronym: LipoaScreen
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Brinck, Associate Professor, Karolinska Institutet
Other Study IDs: K2023-4595
Record Dates: First submitted 2023-11-23; First posted 2023-12-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Dyslipidemias; Hereditary Diseases
Keywords: Lipoprotein(a); Coronary artery disease; Cascade screening; Atherosclerotic cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Genetic Diseases, Inborn; Coronary Artery Disease; Atherosclerosis | interventions — Apolipoproteins A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Index: Patient with atherosclerotic coronary artery disease and a measured plasma lipoprotein(a).
- Biological relative to index: First- or second-degree relative to the index with atherosclerotic coronary artery disease and a measured plasma lipoprotein(a)
  Interventions: Other: measurement of lipoprotein(a)

INTERVENTIONS:
Other: measurement of lipoprotein(a) — Plasma lipoprotein(a) will be measured in the biological relatives group as part of a clinical health care development project
  Groups: Biological relative to index

SUMMARY:
The aim of the current project is to evaluate the penetrance of elevated plasma Lp(a) levels in patients with atherosclerotic coronary artery disease to their first- and second-degree biological relatives based on data from a clinical health care development project.

DETAILED DESCRIPTION:
An elevated plasma level of lipoprotein(a) [Lp(a)] is an independent and causative risk factor for atherosclerotic cardiovascular disease. The Lp(a) plasma level is predominantly genetically determined via a complex hereditary pattern of the LPA gene, and remains relatively constant throughout an individual's entire life cycle. The relationship between plasma Lp(a) and the risk for a cardiovascular event has been shown to be linear.

Cascade screening, i.e. screening of biological relatives of the first detected patient (index) with a disease in a family, is an effective approach to identify and diagnose new patients with hereditary diseases. The method has been shown to be cost-effective for the most common genetically caused dyslipidemia, familial hypercholesterolemia, but the knowledge if cascade screening would be an effective method to screen for elevated plasma Lp(a) is not known.

The aim of the current project is to evaluate the penetrance of elevated plasma Lp(a) levels in patients with atherosclerotic coronary artery disease to their first- and second-degree biological relatives. The study will be based on results from a clinical health care development project in which patients who have had their plasma Lp(a) measured in the clinical routine will be asked to participate in the project. The participating patients invite their relatives to participate in the cascade screening and to measure their plasma Lp(a) levels. Six Swedish hospitals participate in the project and 750 patients with atherosclerotic coronary artery disease be included and divided into three strata according to their plasma Lp(a) level (low <70 nmol/L; intermediate 70-169 nmol/L; high >170 nmol/L). The indexes will in turn invite 1200 first- and second-degree relatives to have their plasma Lp(a) measured.

A scientific evaluation of the health care development project will be performed to study the penetrance of elevated plasma Lp(a) levels in indexes to their relatives.

ELIGIBILITY:
Inclusion Criteria

* participation in the clinical health care development project
* established atherosclerotic coronary artery disease

Exclusion Criteria:

* diagnosis of familial hypercholesterolemia
* chronic kidney disease stadium ≥4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are participating in the clinical health care development project performed at six Swedish hospitals are eligible. Index group consists of patients with atherosclerotic coronary artery disease and a plasma lipoprotein(a) measured in the clinical routine.
  The index invite, according to the health care development project, their first- and second-degree relatives to participate in cascade screening to have their plasma lipoprotein(a) measured .
  Index group, n=750 (n=250 for each lipoprotein(a) strata low, intermediate, high) Relatives group, n=1200 (n=200 for first degree relatives and n=200 for second degree relatives for each of the index lipoprotein(a) strata)
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of elevated plasma lipoprotein(a) between index and first degree relatives | Dataset will be analysed after completion of health care development project (anticipated March 2025)
  Difference in proportion of low, intermediate and high plasma lipoprotein(a) levels between first degree relatives stratified on index patients Lp(a) level (i.e low, intermediate, high)
Difference in proportion of elevated plasma lipoprotein(a) between index and second degree relatives | Dataset will be analysed after completion of health care development project (anticipated March 2025)
  Difference in proportion of low, intermediate and high plasma lipoprotein(a) levels between second degree relatives stratified on index patients Lp(a) level (i.e low, intermediate, high)

SECONDARY OUTCOMES:
Difference in cardiovascular disease burden between index and relatives | Dataset will be analysed after completion of health care development project (anticipated March 2025)
  Difference in prevalence of cardiovascular disease manifestations (coronary artery disease, ischemic stroke, peripheral artery disease) between index and relatives in each of the Lp(a) strata of the index (low, intermediate and high).
  Data on index will be recorded by a health care professional and data on relatives will be self-reported.
Difference in cardiovascular risk factors between index and relatives | Dataset will be analysed after completion of health care development project (anticipated March 2025)
  Difference in prevalence of cardiovascular risk factors (hypertension, diabetes, smoking status) between index and relatives in each of the Lp(a) strata of the index (low, intermediate and high).
  Data on index will be recorded by a health care professional and data on relatives will be self-reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska university hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Due to the General Data Protection Regulation (GDPR) only data on aggregated level will be made available

REFERENCES:
- [Background] Kronenberg F, Mora S, Stroes ESG, Ference BA, Arsenault BJ, Berglund L, Dweck MR, Koschinsky M, Lambert G, Mach F, McNeal CJ, Moriarty PM, Natarajan P, Nordestgaard BG, Parhofer KG, Virani SS, von Eckardstein A, Watts GF, Stock JK, Ray KK, Tokgozoglu LS, Catapano AL. Lipoprotein(a) in atherosclerotic cardiovascular disease and aortic stenosis: a European Atherosclerosis Society consensus statement. Eur Heart J. 2022 Oct 14;43(39):3925-3946. doi: 10.1093/eurheartj/ehac361. PMID 36036785